CLINICAL TRIAL: NCT02318836
Title: Single-Dose Pharmacokinetics and Safety of Oral Lofexidine in Hepatically-Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USWM-LX1-1007; 1R01DA030916 (Other: National Institute on Drug Abuse)
Record Dates: First submitted 2014-07-29; First posted 2014-12-17 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Liver Failure
Keywords: hepatic, hepatic impairment, lofexidine
MeSH Terms: conditions — Liver Failure | interventions — lofexidine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal Hepatic function (Active Comparator)
  Interventions: Drug: Lofexidine Hydrochloride (HCl) tablets
- Mild Hepatic Impairment (Active Comparator): (Child-Pugh score 5-6)
  Interventions: Drug: Lofexidine Hydrochloride (HCl) tablets
- Moderate Hepatic Impairment (Active Comparator): (Child-Pugh score 7-9)
  Interventions: Drug: Lofexidine Hydrochloride (HCl) tablets
- Severe Hepatic Impairment (Active Comparator): (Child-Pugh score 10-15)
  Interventions: Drug: Lofexidine Hydrochloride (HCl) tablets

INTERVENTIONS:
Drug: Lofexidine Hydrochloride (HCl) tablets — Lofexidine HCl tablets (two 200 µg tablets) will be administered orally with 240 mL room temperature tap water as a single 400 µg dose in the morning on Day 1 after a 10 hour overnight fast.

SUMMARY:
This is a Phase 1, open-label, parallel-group, single-dose study of lofexidine in 6 adult subjects with mild hepatic impairment (Child Pugh score of 5 6), 6 adult subjects with moderate hepatic impairment (Child Pugh score 7 9), 6 adult subjects with severe hepatic impairment (Child Pugh score 10 15), and 6 control subjects with normal hepatic function with mean age, body mass index (BMI), and gender distribution targeted to be similar to the impaired hepatic function cohorts.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, parallel-group, single-dose study of lofexidine in 6 adult subjects with mild hepatic impairment (Child Pugh score of 5 6), 6 adult subjects with moderate hepatic impairment (Child Pugh score 7 9), 6 adult subjects with severe hepatic impairment (Child Pugh score 10 15), and 6 control subjects with normal hepatic function with mean age, body mass index (BMI), and gender distribution targeted to be similar to the impaired hepatic function cohorts. Subjects will be confined to an inpatient facility from the evening before dosing to 144 hours after dosing.

Subjects who successfully complete screening will report to the inpatient facility at an appropriate time the evening before study drug administration (Day 1) to ensure a minimum 10 hour fast. The next morning (Day 1) while still fasting, subjects will receive a single, oral dose of 400 µg lofexidine HCl (two 200 µg tablets). Blood samples will be collected for pharmacokinetic (PK) analysis at multiple time points over the next 144 hours (Day 7). Pooled urine samples will be collected at 0 3 hours, 3 6 hours, 6 12 hours, 12 24 hours, 24 48 hours, 48 96 hours, 96 120 hours and 120 144 hours post-dose. Safety will be assessed by recording adverse events (AEs), measuring vital signs (blood pressure and pulse rate) and clinical laboratory tests (chemistry, hematology, and urinalysis), recording 12 lead safety and Holter electrocardiograms (ECGs), and performing physical exams.

ELIGIBILITY:
Inclusion Criteria:

Site will evaluate each subject for criteria in detail, which will include:

1. Between ages of 18 to 65 years at enrollment with a BMI between 19 and 38 kg/m2, inclusive.
2. Subject is eligible to enter the study if:

   * Matched control subject: normal hepatic function and free from other clinically significant illnesses or disease, and medical history, physical examination, laboratory results, and other tests consistent with health, as determined by the Investigator.
   * Subject with mild hepatic impairment: Child-Pugh hepatic dysfunction staging system score of 5-6 Points (Stage A) and medical history, physical examination, laboratory results, and other tests consistent with their hepatic impairment, as determined by the Investigator.
   * Subject with moderate hepatic impairment: Child-Pugh hepatic dysfunction staging system score of 7 9 Points (Stage B) and medical history, physical examination, laboratory results, and other tests consistent with their hepatic impairment, as determined by the Investigator.
   * Subject with severe hepatic impairment: Child-Pugh hepatic dysfunction staging system score of 10-15 Points (Stage C) and medical history, physical examination, laboratory results, and other tests consistent with their hepatic impairment, as determined by the Investigator.

Exclusion Criteria:

Site will evaluate each subject for criteria in detail, which will include:

1. The matched control subject has a history of clinically significant disease, including cardiovascular, gastrointestinal (GI), renal, hepatic, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, or collagen disease or the hepatically-impaired subject has a history of clinically significant disease including cardiovascular, GI, renal, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, or collagen disease.
2. Abnormal cardiovascular exam at Screening, including any of the following:

   * clinically significant abnormal ECG (e.g., second or third degree heart block, uncontrolled arrhythmia, QTcF (Fridericia's correction) interval >450 msec for males and >470 msec for females).
   * heart rate <45 bpm or symptomatic bradycardia;
   * systolic blood pressure <90 mmHg or symptomatic hypotension;
   * blood pressure >160/100 mmHg; or
   * prior history of myocardial infarction.
3. Subjects with hepatic impairment will not be eligible to participate in the study if any of the following exclusion criteria also apply:

   * Significant bleeding diathesis or esophageal bleeding within the last 8 weeks.
   * Evidence of hepatic function deterioration within the last 4 weeks as indicated by liver transaminases, alkaline phosphatase, and gamma-glutamyl transpeptidase or a ≥50% worsening of serum bilirubin or prothrombin time.
   * History of surgical portosystemic shunt.
   * Prothrombin time >18 seconds.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
PK Profile: Cmax, Tmax, AUC, λz, CL/F, T½, CLr, CLd, Ae | pre dose until 144 hours post-dose
  Cmax, Tmax, AUC, λz, CL/F, T½, CLr, CLd, Ae

SECONDARY OUTCOMES:
Adverse events | screening through day 7
Clinical laboratory tests | screening through day 7
  hematology, chemistry, urinalysis
Vital signs | screening through day 7
  blood pressure and pulse
12-lead ECG | screening through day 7
Holter ECG | pre dose through 8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; James Longstreth, PhD, Study Director — USWM, LLC (dba US WorldMeds); Charles Gorodetzky, MD, PhD, Study Director — USWM, LLC (dba US WorldMeds)
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States